CLINICAL TRIAL: NCT00141037
Title: Randomized, Multi-Center Comparative Trial of Tacrolimus w/Steroids and Standard Daclizumab Induction vs a Novel Steroid-Free Tacrolimus Based Immunosuppression Protocol w/ Extended Daclizumab Induction in Pediatric Renal Transplantation
Brief Title: Steroid-Free Versus Steroid-Based Immunosuppression in Pediatric Renal (Kidney) Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Astellas Pharma Inc (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT SNS01
Record Dates: First submitted 2005-08-01; First posted 2005-09-01 (Estimated); Results first posted 2013-07-11 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-10

CONDITIONS: Kidney Diseases; Kidney Transplantation; Kidney Transplant; Renal Transplantation; Renal Transplant
Keywords: Organ Rejection; Corticosteroids; Child; Adolescent; Immunosuppression; Steroids
MeSH Terms: conditions — Kidney Diseases | interventions — Daclizumab; Mycophenolic Acid; Prednisone; Tacrolimus; Ganciclovir; Valganciclovir; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Steroid-Based Immunosuppression (Active Comparator): Subjects will receive prednisone immunosuppression (10 mg/kg peri-operatively followed by 2 mg/kg/day in subjects weighing <40kg and 1.5 mg/kg/day in subjects weighing >40 kg) and proceed with a prednisone taper according to the trial's protocol.
  Interventions: Drug: Daclizumab; Drug: Mycophenolate mofetil (MMF); Drug: Prednisone; Drug: Tacrolimus; Drug: Ganciclovir; Drug: Valganciclovir; Drug: Trimethoprim and sulfamethoxazole
- Steroid-Free Immunosuppression (Experimental): Subjects will receive extended daclizumab induction until the sixth month post-transplant (2 mg/kg pre-transplant followed by 1 mg/kg at weeks 2, 4, 6, 8, 11 and months 4, 5, and 6).
  Interventions: Drug: Daclizumab; Drug: Mycophenolate mofetil (MMF); Drug: Tacrolimus; Drug: Ganciclovir; Drug: Valganciclovir; Drug: Trimethoprim and sulfamethoxazole

INTERVENTIONS:
Drug: Daclizumab — Steroid-Based Immunosuppression(Prednisone) arm: 1 mg/kg pre-transplant followed by 1 mg/kg at weeks 2, 4, 6, and 8 (e.g., standard dose of daclizumab induction until the second month post-transplant)
  Steroid-Free Immunosuppression (Extended daclizumab induction) arm: 2 mg/kg pre-transplant followed by 1 mg/kg at weeks 2, 4, 6, 8, 11, and months 4, 5, and 6 (e.g., extended daclizumab induction until the sixth month post-transplant)
  Other Names: ZENAPAX®; Humanised Anti-Tac Antibody; Ro-24-7375
Drug: Mycophenolate mofetil (MMF) — Intravenous MMF was dosed at 1200 mg/m^2/day in two divided doses preoperatively and for the first 48 hours postoperatively. Oral MMF was dosed at 600 to 900 mg/m^2/day in two divided doses; the dose range allowed for dose titration according to tolerability and side effects of MMF. This regimen was used in both arms.
  Other Names: CellCept®
Drug: Prednisone — Administered as 10 mg/kg peri-operatively followed by 2 mg/kg/day in subjects weighing <40 kg and 1.5 mg/kg/day in subjects weighing >40 kg. The prednisone dosing was tapered as follows: by the end of wks 1, 2, 4,6,12 and 16, dosages were 0.5, 0.4, 0.3, 0.2, 0.15 and 0.1 mg/kg/day, respectively. The prednisone dose of 0.1 mg/kg was achieved by no later than 6 months post-transplant.
  Arms: Steroid-Based Immunosuppression
Drug: Tacrolimus — Taken orally from immediately preoperatively to those>age 5 yrs. (starting dose= 0.1 mg/kg/dose twice daily (BID) for living donor recipients; 0.1 mg/kg/dose daily for deceased donor recipients).Subjects <age 5 yrs. received drug from immediately preoperatively at 0.15 mg/kg/dose BID (two preoperative doses) for living donor recipients and 0.15 mg/kg/dose daily (one preoperative dose) for deceased donor recipients. Postoperatively: 0.07 mg/kg/dose BID w/adjustment to achieve target levels of 12-14 ng/mL (days 0-7), 10-12 ng/mL (wks. 2-8), 7-10 ng/mL (wks. 9-12) &5-7 ng/mL >= 12 wks. Evidence of drug toxicity on any protocol biopsy resulted in a further lowering of the drug target level to 4-6 ng/mL before yr 1 & 3-5 ng/mL after yr 1 post-transplant. This regimen was used in both arms.
  Other Names: Prograf®
Drug: Ganciclovir — Cytomegalovirus (CMV) and Epstein-Barr Virus (EBV) Prophylaxis: All participants will receive intravenous ganciclovir 5 mg/kg/day beginning after transplantation until tolerating oral medications, at which time oral valganciclovir will be initiated and continued for a minimum of 100 days.
  Other Names: Cytovene
Drug: Valganciclovir — Cytomegalovirus (CMV) and Epstein-Barr Virus (EBV) Prophylaxis: All participants will receive intravenous ganciclovir 5 mg/kg/day beginning after transplantation until tolerating oral medications, at which time oral valganciclovir will be initiated and continued for a minimum of 100 days.
  Other Names: Valcyte
Drug: Trimethoprim and sulfamethoxazole — Pneumocystis pneumonia (PCP)/Urinary Tract Infection (UTI) Prophylaxis: Trimethoprim/sulfamethoxazole (Septra®) 2 mg/kg by mouth will be administered daily at bedtime for a minimum period of the first 6 months post-transplant. If unable to tolerate Septra®, inhaled pentamidine (8 mg/kg to a maximum dose of 300 mg monthly) or Dapsone (2 mg/kg PO to a maximum dose of 100 mg/day) may be substituted for a minimum of the first 6 months post-transplant. For UTI prophylaxis, if Septra® is not tolerated, nitrofurantoin (Macrodantin®), 2.5 mg/kg/day, may be given at bedtime up to a maximum dose of 100 mg/day.
  Other Names: Septra®)

SUMMARY:
Over the last 40 years, corticosteroids (steroids) have been an important part of drug regimens used to prevent organ rejection and to maintain the immune health of individuals who have received organ transplants. Unfortunately, the negative physical effects of steroids can be severe, especially in children. The purpose of this study is to determine the safety and effectiveness of a steroid-free treatment regimen for children and adolescents who have received kidney (renal) transplants.

DETAILED DESCRIPTION:
Corticosteroids (steroids) have been a cornerstone of immunosuppressive therapy for kidney (renal) transplantation for over 40 years. However, poor growth and bone loss caused by the use of steroids are devastating to pediatric kidney recipients. The negative physical implications of steroid use also greatly impacts patients' compliance to their prescribed steroid-containing regimens.

The development of a steroid-free regimen for post-transplant pediatric patients is sorely needed. This study will evaluate the safety and efficacy of a steroid-free based treatment regimen in children and adolescents who have received kidney transplants, compared to a standard of care steroid-based regimen. Participants in this study will be pediatric patients with end-stage kidney disease who will undergo kidney transplantation at the start of the study.

Patients will participate in this study for 3 years. Participants will be randomized (1:1) to one of two groups. The study includes 23 study visits over 3 years. A physical exam, medication history, adverse events reporting, blood pressure readings, growth assessment, and blood collection will occur at most visits. At the time of transplantation, participants will have a kidney biopsy. Participants will also undergo cataract screening within 4 months of transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Primary recipient of a kidney transplant
* Meets site-specific transplant criteria
* Panel Reactive Antibody (PRA) of 20% or less
* Willing to use acceptable forms of contraception
* Parent or guardian willing to provide informed consent, if applicable

Exclusion Criteria:

* Previous treatment with steroids within 6 months prior to transplantation
* Received en-bloc kidney or other kidney that does not meet protocol-specified requirements
* Received an organ from an human leukocyte antigen (HLA) identical donor or a non-heart-beating donor
* Received a solid organ other than a kidney
* Received a bone marrow or hematopoietic stem cell transplant
* Received a repeat kidney transplant
* Currently receiving an investigational pharmacologic or biologic agent
* Human Immunodeficiency virus (HIV) infected or infected with another immunodeficiency virus
* Hypersensitivity to murine products or the study drugs or their formulations
* Inability to measure height accurately
* Pregnant or breastfeeding

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 2004-03; Primary Completion 2006-09 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minnie Sarwal, MD, PhD, Study Chair — California Pacific Medical Center; Oscar Salvatierra, MD, Principal Investigator — Pediatric Kidney Transplant Program, Stanford University Medical Center, Stanford Hospital and Clinics
Locations (12):
- United States (12):
  - University of Alabama - Pediatric Nephrology, Birmingham, Alabama
  - Maxine Dunitz Children's Health Center Cedars-Sinai, Los Angeles, California
  - UCLA - Department of Pediatrics, Division of Nephrology, Los Angeles, California
  - Stanford University Medical Center, Lucile Packard Children's Hospital, Palo Alto, California
  - UCSF Children's Hospital, San Francisco, California
  - University of Florida - Pediatric Nephrology, Gainesville, Florida
  - Children's Hospital of New Orleans-Department of Pediatric Nephrology, New Orleans, Louisiana
  - Children's Hospital Boston - Division of Nephrology, Boston, Massachusetts
  - University of Michigan Medical Center, C.S. Mott Children's Hospital- Division of Nephrology & Transplantation, Ann Arbor, Michigan
  - Children's Mercy Hospital - Department of Nephrology, Kansas City, Missouri
  - The Children's Hospital of Philadelphia-Department of Nephrology, Philadelphia, Pennsylvania
  - Children's Hospital & Regional Medical Center - Division of Nephrology, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Background] Cole E, Landsberg D, Russell D, Zaltzman J, Kiberd B, Caravaggio C, Vasquez AR, Halloran P. A pilot study of steroid-free immunosuppression in the prevention of acute rejection in renal allograft recipients. Transplantation. 2001 Sep 15;72(5):845-50. doi: 10.1097/00007890-200109150-00018. PMID 11571448
- [Background] Sarwal MM, Vidhun JR, Alexander SR, Satterwhite T, Millan M, Salvatierra O Jr. Continued superior outcomes with modification and lengthened follow-up of a steroid-avoidance pilot with extended daclizumab induction in pediatric renal transplantation. Transplantation. 2003 Nov 15;76(9):1331-9. doi: 10.1097/01.TP.0000092950.54184.67. PMID 14627912
- [Background] Vidhun JR, Sarwal MM. Corticosteroid avoidance in pediatric renal transplantation. Pediatr Nephrol. 2005 Mar;20(3):418-26. doi: 10.1007/s00467-004-1786-4. Epub 2005 Feb 3. PMID 15690189
- [Background] Vidhun JR, Sarwal MM. Corticosteroid avoidance in pediatric renal transplantation: can it be achieved? Paediatr Drugs. 2004;6(5):273-87. doi: 10.2165/00148581-200406050-00002. PMID 15449967
- [Result] Sarwal MM, Ettenger RB, Dharnidharka V, Benfield M, Mathias R, Portale A, McDonald R, Harmon W, Kershaw D, Vehaskari VM, Kamil E, Baluarte HJ, Warady B, Tang L, Liu J, Li L, Naesens M, Sigdel T, Waskerwitz J, Salvatierra O. Complete steroid avoidance is effective and safe in children with renal transplants: a multicenter randomized trial with three-year follow-up. Am J Transplant. 2012 Oct;12(10):2719-29. doi: 10.1111/j.1600-6143.2012.04145.x. Epub 2012 Jun 13. PMID 22694755
- [Result] Naesens M, Salvatierra O, Benfield M, Ettenger RB, Dharnidharka V, Harmon W, Mathias R, Sarwal MM; SNS01-NIH-CCTPT Multicenter Trial. Subclinical inflammation and chronic renal allograft injury in a randomized trial on steroid avoidance in pediatric kidney transplantation. Am J Transplant. 2012 Oct;12(10):2730-43. doi: 10.1111/j.1600-6143.2012.04144.x. Epub 2012 Jun 13. PMID 22694733
- [Result] Li L, Khatri P, Sigdel TK, Tran T, Ying L, Vitalone MJ, Chen A, Hsieh S, Dai H, Zhang M, Naesens M, Zarkhin V, Sansanwal P, Chen R, Mindrinos M, Xiao W, Benfield M, Ettenger RB, Dharnidharka V, Mathias R, Portale A, McDonald R, Harmon W, Kershaw D, Vehaskari VM, Kamil E, Baluarte HJ, Warady B, Davis R, Butte AJ, Salvatierra O, Sarwal MM. A peripheral blood diagnostic test for acute rejection in renal transplantation. Am J Transplant. 2012 Oct;12(10):2710-8. doi: 10.1111/j.1600-6143.2012.04253.x. PMID 23009139
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- Available data/document: Individual Participant Data Set: SDY132 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY132 — ImmPort study identifier is SDY132
- Available data/document: Study Protocol: SDY132 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY132 — ImmPort study identifier is SDY132
- Available data/document: Study summary, -design,-demographics, -mechanistic assays, -files et al.: SDY132 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY132 — ImmPort study identifier is SDY132

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve pediatric kidney transplantation centers in the United States enrolled 130 subjects (less than 21 years of age) who received a primary kidney transplant from a deceased or living donor. Subject enrollment occurred between March 2004 and July 2006.
Groups:
- Steroid-Free Immunosuppression: Subjects received extended daclizumab induction until the sixth month post-transplant (2 mg/kg pretransplant followed by 1 mg/kg at weeks 2, 4, 6, 8, 11 and months 4, 5, and 6), and maintenance combination tacrolimus and mycophenolate mofetil (MMF) immunosuppression. Anti-viral prophylactic treatment included: 1.) gancyclovir or oral valgancyclovir for at least the first 100 days post-transplantation and 2.) trimethoprim/sulfamethoxazole for a minimum first 6 months post-transplantation. Refer to Registration Assigned Interventions for more details.
- Steroid-Based Immunosuppression: Subjects received prednisone immunosuppression (10 mg/kg peri-operatively followed by 2 mg/kg/day in subjects weighing <40kg and 1.5 mg/kg/day in subjects weighing >40 kg, tapering according to the trial's protocol), standard daclizumab induction until the second month post transplant (1 mg/kg pre-transplant followed by 1 mg/kg at weeks 2, 4, 6, and 8), and maintenance tacrolimus and mycophenolate mofetil (MMF) immunosuppression. Anti-viral prophylactic treatment included: 1.) gancyclovir or oral valgancyclovir for at least the first 100 days post-transplantation and 2.) trimethoprim/sulfamethoxazole for a minimum first 6 months post-transplantation. Refer to Registration Assigned Interventions for more details.
Period: Overall Study
Arm/Group | Steroid-Free Immunosuppression | Steroid-Based Immunosuppression
Started | 60 | 70
Completed | 50 (16 subjects had reduced follow-up) | 52 (8 subjects had reduced follow-up)
Not Completed | 10 | 18
Not completed — Physician Decision | 1 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Other | 0 | 1
Not completed — Moved from area | 1 | 7
Not completed — Graft Failure | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Steroid-Free Immunosuppression | Steroid-Based Immunosuppression | Total
Number analyzed (Participants) | 60 | 70 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.8 (5.4) | 11.9 (6.1) | 11.9 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 28 | 48
  Male | 40 | 42 | 82
Region of Enrollment [Number; unit: participants]
  United States | 60 | 70 | 130

OUTCOME MEASURES:

1. Primary Outcome: The Difference in Linear Growth by Treatment Assignment at 1 Year Post Kidney Transplantation
Description: Standardized Z-scores were computed following a formula using an age- and gender-specific calculation provided by the NHANES III 2000 Growth Data set. The Z-score system expresses anthropometric values of height as several standard deviations (SDs) below (e.g., a negative value) or above (a positive value) the reference mean or median value. In this study the measure was used to test whether there is a difference in the change in height between the treatment groups: Steroid-Based versus Steroid-Free
Time Frame: One year post kidney transplantation procedure
Population: All Enrolled Subjects
Measure: Mean (Standard Deviation); unit: Standard Deviation Score (SDS)
Arm/Group | Steroid-Free Immunosuppression | Steroid-Based Immunosuppression
Number analyzed (Participants) | 60 | 70
Standard Deviation Score (SDS) | 0.37 (0.76) | 0.35 (0.82)
Statistical Analysis 1: Comparison: Steroid-Free Immunosuppression vs Steroid-Based Immunosuppression; The endpoint is assessed using a Wilcoxon nonparametric test and missing values are imputed using the last observation carried forward; Test type: Superiority or Other; p = 0.79, Wilcoxon Nonparametric Test

2. Primary Outcome: Comparison by Treatment Assignment in the Number of Biopsy-Proven Acute Rejections Within 12 Months Post Kidney Transplantation
Description: Biopsy-proven acute renal (kidney) rejection [1, 2].
  1. Diagnosis of acute rejection was made by renal biopsy using the Banff 97 criteria. The Banff 97 diagnostic category for renal allograft biopsies is an international standardized histopathological classification. Acute rejection is defined by a renal biopsy demonstrating a Banff 97 classification of Grade IA or greater, with higher scores indicating more severe rejection[2]
  2. Ref: Racusen LC et al. The Banff 97 working classification of renal allograft pathology. Kidney Int, 55: 713-723, 1999
Time Frame: Up to one year post kidney transplantation procedure
Population: All Enrolled Subjects
Measure: Number (95% Confidence Interval); unit: Rejection Events
Arm/Group | Steroid-Free Immunosuppression | Steroid-Based Immunosuppression
Number analyzed (Participants) | 60 | 70
Rejection Events | 18 [17.85 to 43.21] | 19 [17.20 to 39.10]
Statistical Analysis 1: Comparison: Steroid-Free Immunosuppression vs Steroid-Based Immunosuppression; The difference was analyzed using a Fisher's exact test; Test type: Superiority or Other; p = 0.85, Fisher Exact

ADVERSE EVENTS:
Time Frame: Renal (Kidney) transplantation through end of study
Groups:
- Steroid-Based Immunosuppression: Subjects received prednisone immunosuppression (10 mg/kg peri-operatively followed by 2 mg/kg/day in subjects weighing <40kg and 1.5 mg/kg/day in subjects weighing >40 kg, tapering according to the trial's protocol), standard daclizumab induction until the second month post transplant (1 mg/kg pre-transplant followed by 1 mg/kg at weeks 2, 4, 6, and 8), and maintenance tacrolimus and mycophenolate mofetil (MMF) immunosuppression. Anti-viral prophylactic treatment included: 1.) gancyclovir or oral valgancyclovir for at least the first 100 days post transplantation and 2.) trimethoprim/sulfamethoxazole for a minimum first 6 months post-transplantation. Refer to Registration Assigned Interventions for more details.
Arm/Group | Steroid-Based Immunosuppression | Steroid-Free Immunosuppression
Serious Adverse Events (participants affected / at risk) | 60/70 | 52/60
Other Adverse Events (participants affected / at risk) | 64/70 | 56/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Steroid-Based Immunosuppression (N=70) | Steroid-Free Immunosuppression (N=60)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Congenital nephrotic syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (4)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric outlet obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastro-intestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Difficulty in walking (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 6 (6) | 12 (17)
Graft loss (Immune system disorders) | 3 (3) | 0 (0)
Kidney transplant rejection (Immune system disorders) | 26 (39) | 18 (32)
Transplant rejection (Immune system disorders) | 9 (12) | 6 (6)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Application site abscess (Infections and infestations) | 0 (0) | 1 (1)
BK virus infection (Infections and infestations) | 2 (4) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (2) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Central line infection (Infections and infestations) | 0 (0) | 1 (3)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus hepatitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 3 (3) | 1 (1)
Cytomegalovirus viraemia (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis viral (Infections and infestations) | 0 (0) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 2 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 8 (8) | 3 (3)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (6) | 3 (4)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia primary atypical (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 8 (11) | 7 (10)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 7 (11) | 7 (7)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 3 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Collapse of lung (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Graft dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Treatment noncompliance (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 14 (23) | 20 (41)
Blood potassium increased (Investigations) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Cytomegalovirus antibody positive (Investigations) | 1 (1) | 0 (0)
Cytomegalovirus test positive (Investigations) | 2 (2) | 1 (1)
Drug level below therapeutic (Investigations) | 2 (2) | 1 (1)
Urine output decreased (Investigations) | 2 (3) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 7 (7) | 3 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Schizophrenia (Psychiatric disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Glomerulonephritis focal (Renal and urinary disorders) | 0 (0) | 1 (1)
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 2 (4)
Neurogenic bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 2 (2) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (2) | 1 (3)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Vesicoureteric reflux (Renal and urinary disorders) | 2 (2) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Exposure to communicable disease (Social circumstances) | 1 (1) | 0 (0)
Social problem (Social circumstances) | 1 (1) | 0 (0)
Stent removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Air embolism (Vascular disorders) | 1 (1) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 3 (5) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Lymphocele (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Steroid-Based Immunosuppression (N=70) | Steroid-Free Immunosuppression (N=60)
Anaemia (Blood and lymphatic system disorders) | 21 (21) | 25 (31)
Leukopenia (Blood and lymphatic system disorders) | 12 (22) | 14 (31)
Neutropenia (Blood and lymphatic system disorders) | 21 (27) | 24 (38)
Diarrhoea (Gastrointestinal disorders) | 19 (31) | 18 (26)
Nausea (Gastrointestinal disorders) | 5 (6) | 6 (6)
Vomiting (Gastrointestinal disorders) | 8 (12) | 11 (16)
Pyrexia (General disorders) | 8 (14) | 13 (17)
BK virus infection (Infections and infestations) | 3 (4) | 4 (6)
Cytomegalovirus infection (Infections and infestations) | 6 (7) | 8 (8)
Ear infection (Infections and infestations) | 4 (8) | 6 (7)
Epstein-Barr virus infection (Infections and infestations) | 4 (5) | 6 (7)
Gastroenteritis (Infections and infestations) | 5 (5) | 5 (6)
Otitis media (Infections and infestations) | 8 (9) | 9 (16)
Sinusitis (Infections and infestations) | 8 (14) | 5 (8)
Upper respiratory tract infection (Infections and infestations) | 10 (19) | 20 (28)
Urinary tract infection (Infections and infestations) | 20 (32) | 14 (20)
Incision site complication (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Blood bicarbonate decreased (Investigations) | 4 (6) | 3 (3)
Blood creatinine increased (Investigations) | 6 (10) | 11 (16)
Blood pressure increased (Investigations) | 2 (2) | 6 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 10 (20) | 12 (19)
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 (7) | 6 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 4 (6)
Hypophosphataemia (Metabolism and nutrition disorders) | 12 (12) | 10 (11)
Metabolic acidosis (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Headache (Nervous system disorders) | 7 (8) | 5 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 9 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (7)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 3 (3)
Hypertension (Vascular disorders) | 19 (20) | 14 (15)

LIMITATIONS AND CAVEATS:
1. The results cannot be generalized and daclizumab has since been withdrawn from the United States market (business-related, not due to any safety issues).
2. The study was not powered to definitively evaluate small differences in rejection rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No